CLINICAL TRIAL: NCT05265390
Title: The Effect of Video Informing Adolescents Having Polymerase Chain Reaction (rRT-PCR) Test on Anxiety During the Coronavirus (COVID-19) Pandemic: A Randomized Controlled Study
Brief Title: The Effect of Video Information on Anxiety in Adolescents Having rRT-PCR Test During Corona Virus Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Zühal Artuvan, Specialist Nurse, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Record Dates: First submitted 2022-02-02; First posted 2022-03-03 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Coronavirus
Keywords: Coronavirus; Polymerase Chain Reaction; Adolescent; Anxiety; Information video
MeSH Terms: conditions — Coronavirus Infections; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Anxiety level of the group watching the informational video
  Interventions: Other: Adolescents watching an informational video
- control group (No Intervention): Anxiety level of control group adolescents

INTERVENTIONS:
Other: Adolescents watching an informational video — In the information video; The materials used during the PCR test, how long the process will take, how the sample will be taken, why healthcare professionals wear personal protective equipment, and what adolescents should do are included.
  Arms: intervention group

SUMMARY:
The Polymerase Chain Reaction (rRT-PCR) test is still the gold standard in the diagnosis of coronavirus disease. Health workers apply this procedure in a closed area, wearing personal protective equipment. Adolescents cannot be informed about the invasive procedure and it is difficult to communicate with them. Before the procedure, the effect on anxiety will be investigated by watching an informative video (containing information such as the materials used in the procedure, how long the procedure will take, how the sample will be taken, why healthcare workers wear personal protective equipment) prepared according to the developmental characteristics of the adolescents.

DETAILED DESCRIPTION:
In the coronavirus pandemic, PCR testing is still the gold standard in the diagnosis of the disease. PCR with the right method can increase the sensitivity of the test. Adolescents' anxiety and anxiety levels may increase during invasive procedures such as PCR testing. In addition, in this process, factors such as the uncertainty created by the pandemic, disruption of routines, loss of school and peer social ties, and fear of getting sick bring along many mental disorders. The fact that the tests and treatments for the disease are new and that they are not informed about the procedures to be done cause the anxiety levels of the adolescents to increase. Nurses who treat adolescents with care and personal protective equipment may not be able to communicate verbally, sensorially, eye-to-eye with adolescents, and may have difficulty in conveying their voices and emotions. Likewise, by wearing a mask, it prevents nurses from observing their reactions to the hospital environment and procedures. Video education is one of the most effective ways for nurses to fulfill their educational roles during the epidemic when communication is limited. For this reason, it is very important to inform before the PCR sample collection process with a video prepared in accordance with the developmental stages of the adolescents. The aim of this study is to investigate the effect of the video that adolescents will watch before the procedure on their anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Applying to State Hospital for a PCR test
* Being literate in Turkish
* Not having a hearing or visual impairment, not having a mental disability.
* Not having had a previous PCR test sample taken
* To be in good general condition (clinically)
* Signing the informed consent form (child and parent)

Exclusion Criteria:

* Being illiterate in Turkish
* Hearing or visual impairment, mental disability
* Previous PCR test sample taken
* Absence of parents next to the adolescent
* Those who did not sign the informed consent form (child and parent)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 272 (Actual)
Dates: Start 2022-02-05 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
State Anxiety Inventory Score Form - 1 (STAI FORM -1) | 20 minutes before giving a PCR test sample, the intervention group's State Anxiety Score
  State Anxiety Inventory Score Form - 1. The lowest total score is 20 and the highest total score is 80. A high score indicates a high level of anxiety, and a low score indicates a low level of anxiety.
Trait Anxiety Score Form - 2 (STAI FORM -2) | 20 minutes before giving a PCR test sample, the intervention group's Trait Anxiety Score
  Trait Anxiety Score Form - 2. A total score of 0-19 obtained from the scales indicates no anxiety, a total score of 20-39 indicates mild anxiety, a total score of 40-59 indicates moderate anxiety, and a total score of 60-79 indicates severe anxiety.
Coronavirus Anxiety Scale (CAS) | 20 minutes before giving a PCR test sample, the intervention group's Coronavirus Anxiety Scale Score
  Coronavirus Anxiety Scale - A total score of 9 or more indicates coronavirus-related anxiety.
State Anxiety Inventory Score Form - 1 (STAI FORM -1) | 20 minutes before giving a PCR test sample, the control group's State Anxiety Score
  State Anxiety Inventory Score Form - 1. The lowest total score is 20 and the highest total score is 80. A high score indicates a high level of anxiety, and a low score indicates a low level of anxiety.
Trait Anxiety Score Form - 2 (STAI FORM -2) | 20 minutes before giving a PCR test sample, the control group's Trait Anxiety Score
  Trait Anxiety Score Form - 2. A total score of 0-19 obtained from the scales indicates no anxiety, a total score of 20-39 indicates mild anxiety, a total score of 40-59 indicates moderate anxiety, and a total score of 60-79 indicates severe anxiety.
Coronavirus Anxiety Scale (CAS) | 20 minutes before giving a PCR test sample, the control group's Coronavirus Anxiety Scale Score
  Coronavirus Anxiety Scale - A total score of 9 or more indicates coronavirus-related anxiety.
State Anxiety Inventory Score Form - 1 (STAI FORM -1) | 1 minutes after giving a PCR test sample, the intervention group's State Anxiety Score
  State Anxiety Inventory Score Form - 1. The lowest total score is 20 and the highest total score is 80. A high score indicates a high level of anxiety, and a low score indicates a low level of anxiety.
State Anxiety Inventory Score Form - 1 (STAI FORM -1) | 1 minutes after giving a PCR test sample, the control group's State Anxiety Score
  State Anxiety Inventory Score Form - 1. The lowest total score is 20 and the highest total score is 80. A high score indicates a high level of anxiety, and a low score indicates a low level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Zühal Artuvan, Principal Investigator — Mersin University
Locations (1):
- Mersin Toros Public Hospital, Mersin, Akdeniz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No